CLINICAL TRIAL: NCT00769509
Title: Energy Expenditure Assessment of Preterm Infant With Very Low Birth Weight Fed With Human Milk or Preterm Formula
Brief Title: Energy Expenditure Assessment of Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Maria Elisabeth Lopes Moreira, MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CAAE - 0057.0.008.000-06
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Weight
Keywords: energy expenditure; indirect calorimetry; human milk; preterm formula; premature infant
MeSH Terms: conditions — Body Weight; Premature Birth | interventions — Energy Metabolism

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preterm formula (Experimental): Assessment of energy expenditure of preterm infant during fed with preterm formula
  Interventions: Other: energy expenditure in preterm fed with preterm formula
- human milk with fortifier (Active Comparator): Assessment of energy expenditure by indirect calorimetry during fed with human milk with fortifier
  Interventions: Other: assessment of energy expenditure

INTERVENTIONS:
Other: energy expenditure in preterm fed with preterm formula — Assessment of energy expenditure by indirect calorimetry in preterm infant fed with preterm formula 24 hours before measurements.
  Other Names: energy expenditure
  Arms: preterm formula
Other: assessment of energy expenditure — assessment of energy expenditure in preterm infant during fed with human milk with fortifier
  Other Names: energy expenditure
  Arms: human milk with fortifier

SUMMARY:
The goal of this study is verify if the energy expenditure in preterm infant fed with human milk is different from preterm formula. A randomized, controlled, crossover, double blind clinical trial will be carried out in which the newborn will be its own control. Randomization will be according to the type of diet at the beginning of the study. Half of the participants will be randomly assigned to begin the study using one type of milk (for example, human milk) and later another type of milk (preterm infant formula) and the other half will do the opposite.

DETAILED DESCRIPTION:
Post-natal growth restriction has become a problem yet to be solved and studied in most neonatal units. Newborns with very low birth weight grow at a rate lower than expected, thus culminating with delayed extra-uterine growth, be it in the term assessment, be it at the time of discharge from the hospital, and this makes the search for adequate nutrition a critical issue. Although there are intrinsic risk factors related to prematurity, the nutritional approach of the neonatal unit staff plays a decisive role on the prevalence of malnutrition.

Although the importance of appropriate nutritional management of premature infants has been clearly recognized, the necessary nutrient requirements of most nutrients have not been well established yet and these uncertainties may contribute to a limited intake of nutrients (Hay et al, 1999).

When fresh and extracted mother´s own milk, human milk has been considered the preferred feed for premature newborns, because of its digestibility, balanced chemical composition, capacity to provide immunity and prevention of future diseases (AAP, 2003). In addition, human milk has been associated to lower energy expenditure to be used in comparison with preterm formula, and this may promote the newborn's growth (Lubetzky et al, 2003). However, many of its advantages can be lost when human milk comes from a pool and is pasteurized, and its use has been associated to inadequate weight gain and a nutritional deficit during hospital stay. Thus it is sometimes necessary to use human milk with fortifier or preterm formula, to feed the preterm infant, in order to increase caloric-protein supply and weight gain. Milk formulas for premature babies have currently high caloric density and are better digested, but they do not have the capacity to provide immunity. In face of this problem, several studies are in progress to know and discuss the best nutritional approach for premature newborns during hospital stay. Among the factors that may have an impact on this approach is energy expenditure originated from the type of diet newborns have and on how its caloric constituents (macronutrients) are metabolized.

In face of the aforesaid, the following question remains: Will individually adjusting the caloric density of human and formula milk fed to newborns with very low birth weight actually have any impact on energy expenditure?

2 - OBJECTIVES

2.1 - GENERAL:

- To compare energy expenditure of preterm infants fed with fortified human milk versus preterm infant formula

2.2 - SPECIFIC:

* To analyze the caloric content and macronutrients (fat, protein, and lactose) present in human milk fed to the newborn with very low birth weight at the time of the indirect calorimetry test;
* To analyze the impact of the caloric density of the milk fed to each newborn on energy expenditure;
* To compare the chemical composition of the milks offered to newborns with very low birth weight and their use in energy expenditure
* To analyze the impact of energy substrates on respiratory coefficient;
* To elaborate a pre and post-prandial energy expenditure curve of newborns with very low birth weight for each type of milk fed

  3- MATERIALS AND METHODS

3.1 - Participants: Inclusion criteria:

Newborns admitted to the Intensive Care Unit of Fernandes Figueira Institute with birth weight under 1500g, In order to be included in the study, newborns shall be in room air, with stable growth, without electrolytic unbalance, fed by gavage, with 160/ml/ky/day fluids, alternating human milk and formula for prematurity. Newborns must be tolerating the whole diet, without significant gastric residue (>5% of the total diet).

For ethical reasons, newborns who are exclusively breastfeeding will not be included.

3.1.1 - Exclusion criteria:

Newborns that present the following in their exams shall be excluded: significant gastric residue, signs and symptoms of sepsis, repeated apnea events which required the use of respiratory stimulants.

3.2 - Sample Size Calculation:

Sample size of 25 newborns with very low birth weight was calculated based on the results obtained by Lubetzky et al (2003), considering a 10% difference between energy expenditure of human milk and preterm formula. The level of significance was 95% with a power of the test of 99%. MedCalc software was used in this calculation.

3.3 - Study place

The study will be carried out at the Neonatal Intensive Care Unit of Fernandes Figueira Institute (IFF) / Oswald Cruz Foundation (FIOCRUZ), in Rio de Janeiro - RJ. This research was authorized by the Head of the Neonatology Department of this unit.

3.4 - Main Endpoint

Energy expenditure adjusted by caloric density of milk in both groups measured by open system indirect calorimetry pre and pos feed.

3.5 - Study design

A randomized, controlled, crossover, double blind clinical trial will be carried out in which the newborn will be its own control. Randomization will be according to the type of diet at the beginning of the study. Half of the participants will be randomly assigned to begin the study using one type of milk (for example, human milk) and later another type of milk (preterm infant formula) and the other half will do the opposite.

3.6 Randomization and blinding

Newborns with very low birth weight included in the study will be randomized using a computer generated random numbers table, to initially get human milk and then milk formula or vice-versa. This study will be carried out by researchers whom have been trained to handle all necessary equipment and techniques, as well as to perform the procedures.

Initially the Human Milk Bank will be requested to supply human milk with a caloric value above 65 Kcal/100ml. When it is sent to the Milk Bank for distribution, it will be assessed again by a researcher of the staff, who will be in charge of analyzing the caloric content and macronutrients contained in the milk and of randomization as well. After getting "diet A" for 24 hours, another researcher, who will be "blind", that is, who will not know which diet was given, will perform the indirect calorimetry test, which will be repeated 24 hours after the other type of diet.

The researcher in charge of analyzing the results will also be "blind", that is, he will not know which milk belongs to "diet A" and to "diet B".

3.7 - Study protocol

Energy expenditure assessment

Energy expenditure assessment will be performed by indirect calorimetry, using the Deltatrac II Metabolic Monitor (Datex-Ohmeda, Helsink, Finland. This equipment is based on open circuit principle, which allows measuring oxygen consumption (VO2) and carbon dioxide production (VCO2), using a continuous flow generator.

The indirect calorimetry test will be performed between the 21st and the 28th day of life, period in which the newborn reaches good metabolic stability.

The newborn will be kept inside the incubator, in a thermoneutral zone, with the hood covering its face, without clothing or accessories such as socks, gloves and caps, with clean diapers, in prone position, sleeping or in a state of sleepiness. Temperature will be recorded by a thermometer attached to the infant's skin. The choice of prone position is based on the fact that it is in this position that premature newborns remain quietest, in addition to the many benefits it provides related to the respiratory function. Body movements will be recorded before and during the indirect calorimetry test, following a scale proposed by Thureen (1998), which associates activity and energy expenditure. Measurement will be interrupted when the infants are awake and active or crying.

Deltatrac II has software and a printer connected to it, which provides the average value and standard deviation of the following parameters: baseline energy expenditure, expired CO2 volume, inspired CO2 volume and percentage of use of carbohydrates, proteins and fat, at the end of the test.

The indirect calorimetry test will take place at the following times: 60 minutes before diet administration, 30 minutes during diet through gastroclysis and 90 minutes after diet administration, in a total of 180 minutes.

After having had one type of diet for 24 hours, the indirect calorimetry test will be carried out and right after that the infant will be fed the other type of diet for 24 hours, at the end of which another indirect calorimetry test will be performed. It is necessary to observe a 24 hour washout period to make sure there is no interference of the nutrients from the previous diet, because studies have shown that the thermal effect of food may last for about 18 hours.

The feasibility of obtaining a baseline status of the newborns, that is, a status in which infants remain still for a long period of time, can be assured by the fact that most newborns sleep about 60% of their time and they are in a calm awake state 25% of their time - when metabolism is low. On the other 15% of the time, newborns are either being fed or crying.

Milk analysis In order to assess human milk ingested by the newborn, at the time of the test a 9 ml sample of the milk will be collected - 2ml will be analyzed using creamatocrit and the remaining 7 ml will be sent for qualitative analysis of protein, fat, lactose and total caloric content, dosed by spectrophotometry technique - using INFRARED ANALYSIS (Milko-Scan Minor 104, which has already been validated for human milk analysis. The human milk that will be fed to the newborn, at the time of the test, shall have a caloric value of at least 65 Kcal/100ml.

Formula milk will be calculated using the information provided on the product label, considering volume and dilution and the most commonly used formula is Pré-Nan. The values of preterm formula constituents are Carbohydrate 8,6g/100 ml, protein 2,3g/100 ml, fat 4,2g/100 ml and total kcal is 80 Kcal/100 ml.

Population characteristics

The following anthropometric data will be collected to characterize the population: weight, length, as well as variables related to birth - nutritional status and neonatal practices.

3.8 - Analysis

Data will be entered into a data base created using STATA and the analyses will be performed with STATA software. The analysis of the results will be carried out by variance analysis (ANOVA) for data with normal distribution or Kruskal-Wallis and Wilcoxon for non-parametric data on continuous variables or by chi-square for categoric variables. The regression model will be used for the analysis of association of the variables set considered with the energy expenditure. The choice of variables that will be used in the regression model will be defined based on bivariate analyses. The result will be considered statistically significant if p value is < 0.05.

3.9- Presentation of results

Results will be presented in conformity with the standards suggested by CONSORT, using a flow diagram formed by four phases: selection, assignation, follow-up and analysis, as shown in the scheme below.

4.0- Ethical issues

This project has been approved by the Institutional Review Board for Research with Human Beings of the Fernandes Figueira Institute, under protocol number 0057.0.008.000-06.

The Term of free and informed consent will be requested from the newborn's legal representative, and they will only be included in this research work after the term has been signed.

5 - REFERENCES

American Academic Pediatrics Committee On Nutrition (AAP). Pediatric Nutrition Handbook - 5th Edition. Edited by Ronald E. Kleinman., 2003.

Hay W, Lucas A, Heird WC, Ziegler E, Levin E, Grave GD et al. Workshop Summary: Nutrition of the Extremely Low Birth Weight Infant. Pediatrics 1999; 104 (6):1360-1368.

Lubetzky R, Vaisman N, Mimouni FB, Dollberg S. Energy expenditure in human milk- versus formula-fed preterm infants. J Pediatr 2003; 143(6):750-753.

Thureen PJ, Phillips R, Baron KA. Demarie MP; Hay WWJr. Direct measurement of the energy expenditure of physical activity in preterm infants. J Appl Physiol 1998; 85(1):223-230.

ELIGIBILITY:
Inclusion Criteria:

Premature infant admitted to the Intensive Care Unit of Fernandes Figueira Institute with birth weight under 1500g, adequate for their gestational age, clinically stable, without congenital malformations, nor genetic syndromes confirmed by the geneticist, nor congenital infections confirmed by the physician and lab tests will be eligible for this study, as well as newborn infants who developed intra-ventricular hemorrhage (grades III and IV).

Exclusion Criteria:

Premature infant that present the following in their exams shall be excluded: significant gastric residue, signs and symptoms of sepsis, repeated apnea events which required the use of respiratory stimulants.

Ages: 3 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Energy expenditure adjusted by caloric density of milk in both groups measured by open system indirect calorimetry pre and pos feed With humam milk or preterm formula | from 21 to 28 days of life

SECONDARY OUTCOMES:
weight gain velocity | 2 weeks before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: maria e moreira, MD, Principal Investigator — Oswaldo Cruz Foundation
Locations (1):
- Oswaldo Cruz Foundation, Rio de Janeiro, Brazil